CLINICAL TRIAL: NCT05027347
Title: Detection of Plasma Circulating Tumor DNA in Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Other Study IDs: 79/GCN-HDDD 2021
Record Dates: First submitted 2021-08-25; First posted 2021-08-30 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Circulating Tumor DNA (ctDNA); Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 100 healthy people: 10 ml blood and tissue biopsy were collected from each patient
  Interventions: Diagnostic Test: plasma circulating tumor DNA
- 100 gastric cancer patients: 10 ml blood and tissue biopsy were collected from each patient
  Interventions: Diagnostic Test: plasma circulating tumor DNA

INTERVENTIONS:
Diagnostic Test: plasma circulating tumor DNA — A liquid biopsy assay for identification of tumor derived mutations in plasma of gastric cancer

SUMMARY:
The aim of this study is to develop a protocol for detection of circulating tumor DNA (ctDNA) in plasma of patients with early stages of gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the fifth most common cancer worldwide and the third leading cause of cancer deaths. Earlier detection of GC can dramatically increases the five-year survival rate up to > 90%. The current endoscopy and tissue biopsy remain excessively expensive for middle-income nations, in addition to being fairly invasive, with possible complications. Additionally, most of serum-based biomarkers such as carcinoembryonic antigen (CEA), carbohydrate antigen 19-9 (CA19-9), carbohydrate antigen 72-4 (CA72-4), and carbohydrate antigen 125 (CA125) are not recommended for detection of GC due to the limit of specificity and sensitivity in the early stages of GC. Thus, it is essential to identify new biomarkers for diagnosis of early stages of GC. In this study, the investigators develop an ultradeep massive parallel sequencing (MPS) assay to detect tumor derived mutations (TDM) in plasma of early stages of GC. This study provides proof-of-principle for eventual clinical employment of circulating DNA, via liquid biopsy, for detection of early stages of GC.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients aged 18 years and older
2. Histologically proven stage (I, II and IIIA) gastric adenocarcinoma
3. Naivety to treatment.
4. No known other concomitant cancer diagnosis
5. Signed informed consent

Exclusion Criteria:

1. Pathologically late stage (stage IIIB and IV) or metastatic gastric adenocarcinoma
2. Underwent any type of treatment
3. Unable to undergo biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with early and locally advanced stage (I, II and IIIA) gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and and specificity of our mutation-based assay for detecting early-stage gastric cancer patients | 1 months after collecting blood and specimen
  sensitivity and and specificity of our mutation-based assay for detecting early-stage gastric cancer patients

SECONDARY OUTCOMES:
Limit of detection (LOD): the lowest variant allelic frequency that can be reliably detected | 1 months after collecting blood and specimen
  the lowest variant allelic frequency that can be reliably detected
The concordance rate of mutation results between plasma and tissue biopsy assay | 1 months after collecting blood and specimen
  The concordance rate of mutation results between plasma and tissue biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No